CLINICAL TRIAL: NCT05302284
Title: A Open-Label, Multicenter, Randomised, Controlled Phase 3 Study of RC48-ADC Plus Toripalimab Versus Chemotherapy Alone in Previously Untreated Unresectable Locally Advanced or Metastatic Urothelial Carcinoma With HER2-Expressing
Brief Title: A Study of RC48-ADC Combined With Toripalimab For First-line Treatment of Urothelial Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC48-C016
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Urothelial Carcinoma; HER2-expressing
Keywords: Urothelial Carcinoma; HER2-expressing; RC48; First-Line
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — disitamab vedotin; toripalimab; Gemcitabine; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RC48-ADC + JS001 (Experimental): Participants will receive RC48-ADC + JS001 every 2 weeks (Q2W) until investigator assessed loss of clinical benefit, unacceptable toxicity, investigator or participant decision to withdraw from therapy, or death (whichever occurs first).
  Interventions: Drug: RC48-ADC; Drug: Toripalimab
- Gemcitabine + cisplatin/carboplatin (Active Comparator): Participants will receive Gemcitabine + cisplatin or carboplatin every 3 weeks (Q3W) for maximum 6 weeks or until investigator assessed loss of clinical benefit, unacceptable toxicity, investigator or participant decision to withdraw from therapy, or death (whichever occurs first).
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Drug: Carboplatin

INTERVENTIONS:
Drug: RC48-ADC — 2.0 mg/kg IV every 2 weeks
  Other Names: Disitamab Vedotin
  Arms: RC48-ADC + JS001
Drug: Toripalimab — 3.0 mg/kg IV every 2 weeks
  Other Names: JS001
  Arms: RC48-ADC + JS001
Drug: Gemcitabine — 1000mg/m2 IV infusion on Days 1 and 8 of every 3 week cycle
  Arms: Gemcitabine + cisplatin/carboplatin
Drug: Cisplatin — 70mg/m2 IV infusion on Day 1 of every 3 week cycle
  Arms: Gemcitabine + cisplatin/carboplatin
Drug: Carboplatin — AUC=4.5, IV infusion on Day 1 of every 3 week cycle
  Arms: Gemcitabine + cisplatin/carboplatin

SUMMARY:
This is a Phase 3, Open-Label, Multicenter, Randomised, Controlled Study designed to compare RC48-ADC in Combination With JS001 to Chemotherapy Alone in Previously Untreated HER2-Expressing Unresectable Locally Advanced or Metastatic Urothelial Carcinoma.

DETAILED DESCRIPTION:
This is a Phase 3, Open-Label, Multicenter, Randomised, Controlled Study to evaluate the efficacy and safety of RC48-ADC,a recombinant humanized anti-HER2 monoclonal antibody-Monomethyl auristatin E (MMAE) conjugate, in Combination With JS001,a PD-1 monoclonal antibody, for the treatment of Previously Untreated HER2-Expressing Unresectable Locally Advanced or Metastatic Urothelial Carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Expected survival ≥12 weeks.
* Locally advanced unresectable or metastatic UC with histopathological confirmation, including UC originating from the renal pelvis, ureters, bladder, or urethra.
* Participants must not have received prior systemic therapy for locally advanced or metastatic urothelial carcinoma with the following exceptions:

Participants that received neoadjuvant chemotherapy with recurrence >6 months from completion of therapy are permitted; Participants that received adjuvant chemotherapy following cystectomy with recurrence >6 months from completion of therapy are permitted.

* At least one measurable lesion based on RECIST version 1.1
* HER2-expressing status determined by the central laboratory to be IHC 1+, 2+ or 3+.
* ECOG performance status score: 0 or 1.
* Adequate cardiac, bone marrow, hepatic, renal, and coagulation functions.

Exclusion Criteria:

* Known hypersensitivity to RC48-ADC or Toripalimab or any of its components.
* History of major surgery within 4 weeks of planned start of trial treatment.
* Toxicity from a previous treatment has not returned to Grade 0-1.
* Prior ADCs or PD-1/PD-L1 inhibitor therapy.
* Active central nervous system (CNS) metastases.
* Known active hepatitis B, active hepatitis C, or human immunodeficiency virus (HIV) infection.
* History of other malignancy within the previous 5 years, except for low-risk localized prostate cancer, appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or cancers with a similar curative outcome as those mentioned above.
* Other serious, uncontrolled concomitant diseases that may affect protocol compliance or interpretation of outcomes, including active opportunistic infections or advanced (severe) infections, or uncontrolled diabetes.
* Active autoimmune diseases that require systemic therapy over the past 2 years. Replacement therapies (such as thyroxine, insulin, or physiological replacement of glucocorticoids due to renal or pituitary deficiency) are allowed.
* Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Estimated)
Dates: Start 2022-06-14 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS), evaluated by independent review committee | Up to approximately 3 years
  Progression-free survival (PFS) refers to the time from the date of randomization to the first researcher's evaluation of disease progression or death (calculated by the event that occurred first). The disease progression will be evaluated by independent review committee according to the RECIST 1.1 standard.
Overall survival (OS) | Up to approximately 3 years
  Overall survival (OS) refers to the time from the date of randomization to the date of death of the subject.

SECONDARY OUTCOMES:
Objective remission rate (ORR) | Up to approximately 3 years
  The objective response rate will be mainly analyzed by the independent efficacy evaluation committee according to the RECIST 1.1 standard tumor evaluation (the evaluation by the investigator will also be performed).
Progression-free survival (PFS), evaluated by the investigator | Up to approximately 3 years
  Progression-free survival (PFS) refers to the time from the date of randomization to the first researcher's evaluation of disease progression or death (calculated by the event that occurred first). The disease progression will be evaluated by the researchers according to the RECIST 1.1 standard.
Duration of relief (DOR) | Up to approximately 3 years
  DOR is defined as the time from the first documented objective response (CR or PR) to the first documented disease progression or death
Disease control rate (DCR) | Up to approximately 3 years
  Disease control rate (DCR) is defined as cases where objective remission (assessed as complete remission or partial remission according to RECIST 1.1 standard) or stable disease during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Na Su, PhD, Study Director — RemeGen Co., Ltd.
Locations (2):
- China (2):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing

REFERENCES:
- [Derived] Sheng X, Zeng G, Zhang C, Zhang Q, Bian J, Niu H, Li J, Shi Y, Yao K, Hu B, Liu Z, Liao H, Yu Z, Jin B, Zhao P, Yang T, Liu X, Qin Y, Xue X, Gou X, Huang J, Gu J, Qi X, Zhang L, Ma G, Liu B, Fang J, Jiang S, He Z, Zhou A, Guo J; RC48-C016 Trial Investigators. Disitamab Vedotin plus Toripalimab in HER2-Expressing Advanced Urothelial Cancer. N Engl J Med. 2025 Dec 11;393(23):2324-2337. doi: 10.1056/NEJMoa2511648. Epub 2025 Oct 19. PMID 41124210